CLINICAL TRIAL: NCT00699673
Title: Evaluation of the Brain Natriuretic Peptide as a Predictor of Morbidity and Mortality in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 3910
Record Dates: First submitted 2008-06-10; First posted 2008-06-18 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease; Valvular Disease
Keywords: Brain natriuretic peptide; EuroScore; Cardiac surgery; Cardiopulmonary bypass; Coronary artery disease; Valvular disease; Risk stratification in cardiac surgery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: The purpose of the present study is to assess if perioperative variation of Brain Natriuretic Peptide (BNP) levels is a predictor of mortality and morbidity after cardiac surgery.Material and Methods: 500 consecutive patients will be enrolled prospectively in this study before cardiac surgery under cardiopulmonary bypass. BNP levels will be measured prior to surgery and at postoperative day 1. Variations of BNP levels will be analyzed to determine if it is a predictor of mortality and morbidity after cardiac surgery. This dynamic evaluation will be compared to other tools of risk stratification in cardiac surgery as the EuroScore. All patients will be followed 3 years after the procedure.

Hypothesis: Perioperative BNP variations may be more sensitive than pre- or postoperative BNP levels alone. Furthermore the perioperative homeostasis will be measured to assess its impact on BNP secretion during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patient who need cardiac surgery
* Age > 18 years

Exclusion Criteria:

* Patient on mechanic ventilation before surgery
* Aortic dissection-Congenital disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who need cardiac surgery and age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
BNP levels; hospital and long-term morbidity and mortality | BNP levels prior to surgery and at postoperative day 1; Hospital and long-term morbidity and mortality (1, 2 and 3 years)

SECONDARY OUTCOMES:
EuroScoreCardiac markers; inflammation markers; echocardiography | EuroScoreCardiac markers at day 1, 2, 5; Inflammation markers at day 1, 2, 5; Echocardiography (day 5, and 1, 2 and 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Michel KINDO, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Chirurgie Cardio-Vasculaire au NHC, Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Derived] Kindo M, Minh TH, Perrier S, Petit-Eisenmann H, Bentz J, Cristinar M, Ajob G, Collange O, Mazzucotelli JP. Impact of prosthesis-patient mismatch on early haemodynamic status after aortic valve replacement. Interact Cardiovasc Thorac Surg. 2017 Jan;24(1):48-54. doi: 10.1093/icvts/ivw303. Epub 2016 Sep 13. PMID 27624355